CLINICAL TRIAL: NCT00503074
Title: Starting Healthy Staying Healthy Pilot Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: Seattle Children's Hospital (Other)
Responsible Party: Frederick J. Zimmerman, Associate Professor, University of Washington
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 07-6609-J01
Record Dates: First submitted 2007-07-16; First posted 2007-07-18 (Estimated); Last update posted 2009-11-20 (Estimated); Status verified 2009-11

CONDITIONS: Obesity
Keywords: Diet, reducing; Television; Child Behavior
MeSH Terms: conditions — Obesity; Child Behavior | interventions — Safety

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Parents receive tailored health-behavior change messages designed to reduce their child's exposure to televised food commercials. Intervention is delivered by a case manager, by a website, and by periodic newsletters.
  Interventions: Behavioral: TV modification
- Control (Active Comparator): Parents of children ages 2-5 receive behavioral-change counseling around toddler & preschooler safety and injury prevention.
  Interventions: Behavioral: safety and injury prevention

INTERVENTIONS:
Behavioral: TV modification — Parents receive a health behavior-change intervention consisting of 1 in-person visit from a case manager, followed by phone and e-mail contact at least monthly. The intervention is designed to promote healthy TV viewing, including viewing fewer commercials, by the target child aged 2-5 years old, and uses health behavior change theory and social cognitive theory.
  Arms: 1
Behavioral: safety and injury prevention — Parents receive behavior-change counseling around toddler and preschooler safety and injury prevention.
  Arms: Control

SUMMARY:
The purpose of this study is to determine whether a reduction in toddlers' and preschoolers' exposure to television advertising leads to a change in their diet.

DETAILED DESCRIPTION:
TV viewing is among the most significant features of childhood. In the past generation or two, new technologies have made media viewing more ubiquitous and frequent: 30% of children eat regularly in front of TV, one-third under 6 have TVs in their bedrooms, and 30% make TV part of bedtime routines. By the age of 2 years, 90% of children watch TV or videos regularly. Among those who watch, average viewing is 1.5 hours daily by age 2.

Yet the effects of this early viewing are poorly understood. In this study, we focus on children's diet, because children's food preferences have been shown to be easily influenced by advertising, and children's non-educational programming is heavy with advertising for poor nutritional-quality foods.

We will recruit 70 families with children ages 24-30 months and randomize them to either a television-minimization intervention (the intervention arm) or a toddler safety and injury prevention arm (the control arm). A case manager will actively work with the intervention arm participants to strategize ways of minimizing their media exposure. In addition, families in the intervention arm will get access both to a study website and to a monthly newsletter. The website and newsletter will inform participants of the potential hazards of early media exposure, and will offer tips for alternative activities and strategies for keeping children occupied while the parent gets a much-needed break. The control arm will have no case manager, but will have access to a website and newsletter that will emphasize toddler safety and injury-prevention themes. At the conclusion of the 4-month trial, we will assess (a) whether the study participants regularly accessed their respective websites; (b) whether the intervention-arm participants have different beliefs and attitudes about television for toddlers; and (c) whether fewer intervention-arm children watch TV compared to control-arm infants.

The comparison group will receive a similar intervention, except that it will not mention television viewing, and will instead focus on toddler and preschooler safety and injury-prevention topics, such as the appropriate use of car seats, smoke detectors, hot water heater temperature, safe gun storage, and other similar topics.

ELIGIBILITY:
Inclusion Criteria:

* Must watch at least 1.5 hours of television a day on average
* Must speak English at home
* Residence in or near Seattle

Exclusion Criteria:

* Developmental delay

Ages: 2 Years to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 70 (Estimated)
Dates: Start 2007-07; Primary Completion 2008-02 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Consumption of foods frequently advertised on television (sugary cereals, sugary beverages, candy, fast food, salty snacks) | at conclusion of trial and 6 months post-intervention

CONTACTS AND LOCATIONS:
Overall Officials: Frederick J Zimmerman, Ph.D., Principal Investigator — University of Washington
Locations (1):
- Child Health Institute, University of Washington, Seattle, Washington, United States

REFERENCES:
- [Derived] Zimmerman FJ, Ortiz SE, Christakis DA, Elkun D. The value of social-cognitive theory to reducing preschool TV viewing: a pilot randomized trial. Prev Med. 2012 Mar-Apr;54(3-4):212-8. doi: 10.1016/j.ypmed.2012.02.004. Epub 2012 Feb 14. PMID 22349644